CLINICAL TRIAL: NCT04934293
Title: Virtual Reality for Children in Radiotherapy (REVER)
Acronym: REVER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020/04
Record Dates: First submitted 2021-06-14; First posted 2021-06-22 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Virtual Reality; Proton Therapy; Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Open-label, monocentric, randomized (1:1), stratified, cross-group cohort study (cross-over), comparing the use of the virtual reality headset from the first session (Arm A) versus the use of the virtual reality from the sixth session (Arm B) of proton therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A_ first with RV then without (Experimental): Use of the virtual reality headset from the first week of proton therapy
  Interventions: Procedure: Virtual reality
- Arm B- first without RV than with (Experimental): Use of the virtual reality headset from the second week of proton therapy
  Interventions: Procedure: Virtual reality

INTERVENTIONS:
Procedure: Virtual reality — Before proton therapy, virtual reality sessions will be performed.

SUMMARY:
For a young patient, the conditions of proton therapy treatment can be stressful. Adjusting the environment can be a source of avoiding this physical and psychological discomfort impacting the quality of treatment.

A fixed, long, uncomfortable position is the main cause of stress, already present due to the cancerous therapeutic course. It extends the positioning time. For the patient and the optimization of his treatment, solutions must be sought.

Relaxation in virtual reality is efficient, simple and non-medicinal and could reduce stress in children and allow irradiation in very good conditions.

We will assess the effectiveness of the virtual reality session using objective (placement time, helmet tolerance) and subjective (perceived anxiety via a dedicated questionnaire) criteria. This is the first pediatric virtual reality study, supported by the French Group of Pediatric Radiotherapists, to reduce anxiety in radiotherapy.

Multiple benefits from this pilot study are expected, such as improved reception conditions, treatment parameters and better acceptance of proton therapy sessions.

DETAILED DESCRIPTION:
The treatment of certain pediatric cancers requires irradiation. These treatments are stressful in children because it is necessary to keep a fixed position that is often uncomfortable. The more the stress increases, the longer the positioning, which again generates stress making the treatment position more and more uncomfortable. This irradiation can be carried out by various conventional techniques, tomotherapy, proton therapy. In all cases, the precise positioning, essential for the successful completion of the treatment, under the treatment machine is an iterative process, requiring long and tedious checks. This positioning step on the treatment table takes about 15 minutes, but depending on the technical difficulty can be extended up to 45 minutes in the most complex cases and depending on the patient's apprehension. This positioning is then checked by placement verification images.

At the Antoine LACASSAGNE Center, the investigators have a new generation proton therapy device. This device allows radiotherapy doses to be delivered extremely precisely, subject to very rigorous positioning, and is therefore particularly suitable for pediatric treatment by protecting organs near the radiation. In addition, proton therapy requires longer sessions than conventional radiotherapy; which generates even more anxiety for the children for whom it is the treatment of choice. Non-drug solutions to reduce this stress are therefore necessary to allow the irradiation to be carried out under optimal conditions in order to ensure the effectiveness and safety of the treatment. In this context, virtual reality (VR) headsets, using relaxation techniques in virtual reality or digital sedation, are presented as a simple solution to reduce the anxiety of children regarding the treatment and would therefore be tested mainly on this modality.

To allow us to assess the effectiveness of this technique on anxiety, the investigators will therefore measure the positioning time necessary before carrying out a treatment session and its reduction via its impact on perceived anxiety thanks to a dedicated questionnaire.

The strength of our study is that it uses simple and reproductive measurement systems such as the measurement of placement time and a validated anxiety scale during Marie POURCHET's science thesis. This is the easy EVAN (Anxiety Assessment) scale adapted to several age groups and developed in pediatric wards.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated at the Antoine LACASSAGNE Center for treatment by proton therapy
* Age ≥ 7 years old and ≤ 18 years old
* Patient, and parents for minor children, having read the information notice and signed the informed consent,
* Patient with social security coverage.

Exclusion Criteria:

* Age < 7 years old and > 18 years old,
* Patient under general anesthesia,
* Patient suffering from wounds or infections in the head, deemed incompatible with the use of the helmet by the investigator,
* Patient suffering from respiratory problems,
* Patient suffering from a high level of claustrophobia,
* Patient followed for a psychiatric pathology,
* Patient suffering from unbalanced epilepsy,
* Patient suffering from visual (binocular vision) and / or hearing disorders preventing the use of virtual reality,
* Patient whose head circumference is insufficient for the use of the helmet, deemed incompatible with the use of the helmet by the investigator,
* Patient treated by radio chemotherapy.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Estimated)
Dates: Start 2021-08-02 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Impact of sedation | 2 weeks
  The first co-primary endpoint of the study is the measurement of the duration of positioning before irradiation; from installation on the table in a lying position to return to the console to start the irradiation (imaging time included). The measurement of this parameter will make it possible to compare the difference in positioning time with and without digital sedation during the first 5 proton therapy sessions.
Benefits of using the virtual reality headset from the first proton therapy session | 2 weeks
  The second co-primary endpoint of the study is the comparison of the difference in positioning time over the first 10 sessions when the virtual reality headset is used from the first session or when it is used from the sixth proton therapy session

SECONDARY OUTCOMES:
Change in anxiety before irradiation | 2 weeks
  The measurement before each irradiation session of the anxiety in the child using the EVAN questionnaire. Measuring this parameter will assess: the difference in anxiety before irradiation with and without digital sedation
The tolerance of the virtual reality procedure | 2 weeks
  The evaluation of the tolerance of the virtual reality procedure before the proton therapy session by recording the appearance and intensity of an adverse event during the digital sedation session, mainly headache, drowsiness, dizziness, anxiety, creation of false memories, dizziness, eye or muscle twitching or loss of consciousness on light stimulation, eye strain, impaired vision, disorientation, imbalance, coordination disorder, panic or anxiety attack, nausea, vomiting. The toxicities will be reported in the evaluation grid.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: No